CLINICAL TRIAL: NCT01139996
Title: A Randomized Double Blinded Placebo Controlled Trial Of Transdermal Clonidine for Adjuvant Sedation in Ventilated Trauma Patients Experiencing Delirium
Brief Title: Use of Transdermal Clonidine in Trauma Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty in enrolling participants
Sponsor: Memorial Health University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MHUMC-2010-04-02
Record Dates: First submitted 2010-06-07; First posted 2010-06-09 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium | interventions — Clonidine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transdermal Clonidine/Oral Clonidine (Experimental): An oral loading dose of Clonidine 0.3 mg and placement of a Clonidine Transdermal system at a dose of 0.3 mg/day (Catapres TTS-3), with patch overlay, followed by a final dose of Clonidine 0.3 mg after 12 hours
  Interventions: Drug: Clonidine
- Comparator (Placebo Comparator): Placebo group will receive a placebo oral tablet and the overlay patch only and in 12 hours they will receive a second and final placebo tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clonidine — An oral loading dose of Clonidine 0.3 mg and placement of Clonidine Transdermal system at a dose of 0.3-mg/day (Catapres TTS-3), with patch overlay, followed by a final dose of Clonidine 0.3mg after 12 hours
  Arms: Transdermal Clonidine/Oral Clonidine
Drug: Placebo — A placebo oral tablet and the overlay patch only and in 12 hours they will receive a second and final tablet
  Arms: Comparator

SUMMARY:
This study will attempt to learn how to better treat trauma patients with delirium who are on a breathing machine. Delirium, also known as acute, temporary brain dysfunction, is a common reason why ventilated patients can not be weaned from the breathing machine even though their lungs may be healthy enough to breathe without the machine. The study hopes to show that by decreasing the patient's delirium it will lead to quicker weaning from the breathing machine and possibly a quicker overall recovery as well. Patients enrolled in this study will be treated with Clonidine or placebo. Clonidine is a drug that produces significant calming effects, decreases anxiety, and reduces pain, but with a lower incidence of delirium than other medications used in the ICU for this purpose. Clonidine is not approved by the Federal Food and Drug Administration for treatment of delirium, but is commonly used for this purpose.

DETAILED DESCRIPTION:
Obtaining the appropriate level of sedation and analgesia in severely injured trauma patients admitted to the intensive care unit (ICU) can be challenging due to the diversity of injuries as well as the breadth of comorbidities present in this population. Clonidine may be a useful adjuvant to traditional analgesics such as opioids and sedatives such as benzodiazepines and propofol. Ventilator dependent trauma patients frequently fail extubation trials secondary to inappropriate sedation, inadequate analgesia or undertreated delirium. Patients that fail extubation for these reasons have a potentially preventable prolonged ventilator, ICU and hospital course. Ventilated trauma patients that meet criteria for our institution's SBT protocol and have the diagnosis of delirium will be considered for the trial if they have a documented failed SBT. We hypothesize treatment of this patient population with transdermal Clonidine will decrease delirium in trauma patients during their ICU stay. Patients enrolled in the treatment group will receive an oral loading dose of Clonidine 0.3 mg and placement of a Clonidine Transdermal system at a dose of 0.3-mg/day (Catapres TTS-3) covered by a patch overlay. In 12 hours the patient will receive a second and final dose of Clonidine 0.3 mg. The placebo group will receive a placebo oral tablet and the overlay patch only and in 12 hours they will receive a second and final placebo tablet. A total of 120 patients will be enrolled, 60 patients in each group. All patients will complete the study at end of Day 14 or upon discharge from the hospital, whichever comes sooner. Ventilator times will be measured in each group as well as the prevalence of delirium by the amount of positive CAM-ICU scores over the course of the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Ventilated male or female trauma patient 18 years of age or older admitted to the ICU >24 hours
2. Patient must meet minimal medical criteria for potential extubation (meet criteria for being placed on spontaneous breathing trials per established MUMC SBT protocol)
3. Patients must exhibit delirium as assessed by the CAM-ICU assessment tool
4. Patient must be declared stable from a neurologic, respiratory and cardiovascular standpoint to receive clonidine by the attending MD
5. Consent must be obtained prior to any study procedures

Exclusion Criteria:

1. Patient < 18 years old
2. Bradycardia (HR < 60)
3. Presence of active pacemaker
4. Hypotensive (<90/60)or active treatment of hypotension with vasoactive medications
5. Patient actively being treated with Clonidine or dexmedetomidine
6. Presence of allergy to Clonidine
7. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-05; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Memorial Health University Medical Center, Savannah, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Transdermal Clonidine/Oral Clonidine | Comparator
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: baseline data were not collected
Groups:
- Total: Total of all reporting groups
Arm/Group | Transdermal Clonidine/Oral Clonidine | Comparator | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Continuous
Sex: Female, Male
Adjuvant Sedation and Anxiolysis

OUTCOME MEASURES:

1. Primary Outcome: Duration of Mechanical Ventilation Following Administration of the First Dose of Clonidine or Placebo
Description: data were not collected
Time Frame: 2 or more years
Population: data were not collected
Arm/Group | Transdermal Clonidine/Oral Clonidine | Comparator
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Incidence and Duration in Hours of Delirium Currently Used
Description: As assessed by the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) score Data were not collected
Time Frame: 2 or more years
Reporting Status: Not Posted

3. Secondary Outcome: Time to Pass First SBT Following Administration of the First Dose of Clonidine or Placebo
Description: Hours. data were not collected
Time Frame: 2 or more years
Reporting Status: Not Posted

4. Secondary Outcome: Mean Incidence and Duration of Delirium
Description: As assessed by daily CAM score currently used. data were not collected
Time Frame: 2 or more years
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: data were not collected
Arm/Group | Transdermal Clonidine/Oral Clonidine | Comparator
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes